CLINICAL TRIAL: NCT00598702
Title: A Phase III Multi-Center, Open-Label, Prospective, Repeated Dose, Multi-Day Study of the Safety & Efficacy of Intravenous Acetaminophen in Pediatric Inpatients.
Brief Title: Study of the Safety & Efficacy of Intravenous Acetaminophen in Pediatric Inpatients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPI-APA-352
Record Dates: First submitted 2008-01-09; First posted 2008-01-22 (Estimated); Results first posted 2011-01-06 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Pain; Fever
MeSH Terms: conditions — Pain; Fever | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV Acetaminophen (Experimental): 40 to 75 mg/kg/day every 4 to 6 hours
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen — Target is 1 to 7 days of therapy with intravenous (IV) Acetaminophen (IV APAP) at a dose of 40 to 75 mg/kg body weight/day administered as an IV infusion (or by syringe pump) over 15 minutes and given every 4 to 6 hours as a scheduled dose
  Other Names: IV APAP; APAP

SUMMARY:
Intravenous acetaminophen (IVAPAP) is safe in repeated dose, multi-day clinical use when administered at a daily dose of 40 to 75 mg/kg body weight

DETAILED DESCRIPTION:
To assess the safety of intravenous acetaminophen (IV APAP) when used over one or more days for the treatment of acute pain or fever in pediatric (neonates, infants, children and adolescents) inpatients who are unable to take anything by mouth (NPO), require or would benefit from IV treatment, or are willing and able to stay on IVAPAP therapy for 1 to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* The Subject's Parent or Guardian must provide written informed consent, with Subject assent where appropriate, prior to the Subject's participation in the Study.
* Be less than 17 years of age and older than 37 weeks post conception
* Anticipated by the Investigator to require multi-day (minimum of one day) use of intravenous (IV) treatment either because of a having a status of nothing by mouth (NPO) or a medical condition that makes oral intake difficult or be willing to undergo at least 5 days of treatment with IV acetaminophen for the treatment of pain or fever
* Have the ability to read and understand the Study procedures and have the ability to communicate meaningfully with the Study Investigator and staff (if the Subject is of preverbal age or cannot read or communicate meaningfully, then the Subject's Parent or Guardian must meet this criterion)
* If a female of child bearing potential, have a negative pregnancy test

Exclusion Criteria:

* Has significant medical disease(s), laboratory abnormalities or condition(s) that in the Investigator's judgment could compromise the Subject's welfare, ability to communicate with the Study staff, complete Study activities, or would otherwise contraindicate Study participation
* Has known hypersensitivity or contraindication to receiving IV acetaminophen or the inactive ingredients (excipients) of IV acetaminophen
* Has impaired liver function, e.g. Alanine aminotransferase (ALT) greater than or equal to 3 times the upper limit of normal (ULN), bilirubin greater than or equal to 3 times ULN, known active hepatic disease (e.g., hepatitis), evidence of clinically significant chronic liver disease or other condition affecting the liver (e.g., alcoholism as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), cirrhosis, or chronic hepatitis) that may suggest the potential for an increased susceptibility to hepatic toxicity with IV acetaminophen exposure
* Has participated in an interventional clinical Study (investigational or marketed product) within 30 days of Study entry

Ages: 37 Weeks to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Lucile Salter Packard Children's Hospital at Stanford, Stanford, California
  - Alfred Dupont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Ann Arbor, Ann Arbor, Michigan
  - University of Missouri, Columbia, Missouri
  - Hospital for Special Surgery, New York, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Houston Neonatal-Perinatal Physicians, Bellaire, Texas
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-center study conducted in the United States from 19 Mar 2008 - 24Dec 2008
Pre-assignment Details: No subjects were entered into the "Infants (29 days to 1 year old): IV APAP 6.7 - 12.5 mg/kg q4h" group
Groups:
- Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h: Neonates 28 days or less who were administered 10 -15 mg/kg body weight intravenous acetaminophen solution every 8 hours
- Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h: Infants 29 days to 1 year old who were administered 10 -15 mg/kg body weight intravenous acetaminophen solution every 6 hours
- Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h: Children 2 to < 12 years old who were administered 6.7 -12.5 mg/kg body weight intravenous acetaminophen solution every 4 hours
- Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h: Children 2 to < 12 years old who were administered 10 -15 mg/kg body weight intravenous acetaminophen solution every 6 hours
- Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h: Adolescents 12 to <= 16 years old who were administered 6.7 -12.5 mg/kg body weight intravenous acetaminophen solution every 4 hours
- Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h: Adolescents 12 to <= 16 years old who were administered 10 - 15 mg/kg body weight intravenous acetaminophen solution every 6 hours
- Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h: Infants 12 to < 24 months who were administered 6.7 -12.5 mg/kg body weight intravenous acetaminophen solution every 4 hours
- Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h: Infants 12 to < 24 months who were administered 10 - 15mg/kg body weight intravenous acetaminophen solution every 6 hours
Period: Overall Study
Arm/Group | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h
Started | 1 | 3 | 7 | 33 | 9 | 42 | 1 | 4
Completed | 1 (Completed treatment period per requirements of protocol version under which the subject enrolled.) | 1 (Completed treatment period per requirements of protocol version under which the subject enrolled.) | 5 (Completed treatment period per requirements of protocol version under which the subject enrolled.) | 25 (Completed treatment period per requirements of protocol version under which the subject enrolled.) | 6 (Completed treatment period per requirements of protocol version under which the subject enrolled.) | 30 (Completed treatment period per requirements of protocol version under which the subject enrolled.) | 0 (Completed treatment period per requirements of protocol version under which the subject enrolled.) | 4 (Completed treatment period per requirements of protocol version under which the subject enrolled.)
Not Completed | 0 | 2 | 2 | 8 | 3 | 12 | 1 | 0
Not completed — Other | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Early discharge from hospital | 0 | 0 | 2 | 5 | 0 | 10 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Dose limiting toxicity | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h | Total
Number analyzed (Participants) | 1 | 3 | 7 | 33 | 9 | 42 | 1 | 4 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 7 | 33 | 9 | 42 | 1 | 4 | 100
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 5 | 17 | 6 | 29 | 0 | 3 | 62
  Male | 1 | 1 | 2 | 16 | 3 | 13 | 1 | 1 | 38

OUTCOME MEASURES:

1. Secondary Outcome: Subject's (Parent/Guardian) Global Evaluation of Study Treatment
Description: Subject's (parent/guardian) was asked to evaluate the overall study treatment using a 4-point categorical evaluation scale (0= poor, 1= fair, 2=good, 3= excellent).
Time Frame: Day 0 to Day 5, Day 7 or Early Termination from study
Population: All analysis will be carried out using the safety population, defined as all subjects who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h
Number analyzed (Participants) | 1 | 3 | 7 | 33 | 9 | 42 | 1 | 4
participants
  Poor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fair | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
  Good | 0 | 3 | 1 | 11 | 3 | 17 | 0 | 1
  Excellent | 1 | 0 | 6 | 17 | 5 | 23 | 1 | 2
  Missing | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Subjects Reporting at Least One Treatment Emergent Adverse Event (TEAE)
Description: A TEAE is defined as an adverse event that starts on or after the start of study medication.
Time Frame: First dose to end of treatment period
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h
Number analyzed (Participants) | 1 | 3 | 7 | 33 | 9 | 42 | 1 | 4
Subjects | 1 | 1 | 5 | 25 | 9 | 35 | 0 | 2

3. Secondary Outcome: Physician's Global Assessment of Study Treatment
Description: Physicians were asked to evaluate the overall study treatment using a 4-point categorical evaluation scale (0= poor, 1= fair,2=good, 3= excellent).
Time Frame: End of study or Early Termination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h
Number analyzed (Participants) | 1 | 3 | 7 | 33 | 9 | 42 | 1 | 4
participants
  Poor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fair | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Good | 0 | 2 | 1 | 15 | 4 | 16 | 0 | 1
  Excellent | 1 | 1 | 6 | 13 | 5 | 25 | 1 | 2
  Missing | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Subjects Reporting at Least One Serious Treatment Emergent Adverse Event
Description: A Serious Treatment Emergent Adverse Event is defined as any untoward medical occurrence at any dose of IV APAP that;
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or causes prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * is an important medical event
Time Frame: First dose to 30 days after last dose
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h
Number analyzed (Participants) | 1 | 3 | 7 | 33 | 9 | 42 | 1 | 4
Subjects | 1 | 1 | 0 | 13 | 2 | 3 | 0 | 1

ADVERSE EVENTS:
Time Frame: Non-serious treatment emergent adverse events (TEAEs) were collected from the initiation of treatment with study medication to the end of the patient's treatment period.
Description: Serious adverse events (SAEs) were collected from the initiation of study medication through 30 days of the last dose of study drug.
Arm/Group | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/3 | 0/7 | 13/33 | 2/9 | 3/42 | 0/1 | 1/4
Other Adverse Events (participants affected / at risk) | 1/1 | 1/3 | 5/7 | 24/33 | 9/9 | 33/42 | 0/1 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h (N=1) | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h (N=3) | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h (N=7) | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h (N=33) | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h (N=9) | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h (N=42) | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h (N=1) | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h (N=4)
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 (0) | 0 (0) | 0 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 (0) | 0 (0) | 0 | 0
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 (0) | 0 (0) | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Congenital Megacolon (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Exacerbation of Hirschsprung's Disease
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter-Related Complication (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Accidental dislodgement of suprapubic cathether
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neonates (<= 28 Days Old): IV APAP 10 - 15 mg/kg q8h (N=1) | Infants (29 Days to 1 Year Old): IV APAP 10 - 15 mg/kg q6h (N=3) | Children (2 to < 12 Years Old): IV APAP 6.7 - 12.5 mg/kg q4h (N=7) | Children (2 to < 12 Years Old): IV APAP 10 - 15 mg/kg q6h (N=33) | Adolescents (12 to <= 16 Years): IV APAP 6.7 - 12.5 mg/kg q4h (N=9) | Adolescents (12 to <= 16 Years Old): IV APAP 10 - 15 mg/kg q6h (N=42) | Infants (12 to < 24 Months): IV APAP 6.7 - 12.5 mg/kg q4h (N=1) | Infants (12 to < 24 Months): IV APAP 10 - 15 mg/kg q6h (N=4)
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 11 | 2 | 10 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 4 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Laryngotracheal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 6 | 5 | 17 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 5 | 4 | 4 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 7 | 0 | 3 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum culture positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 7 | 4 | 10 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Infusion Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-Glutamyltransferase (GGT) Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound Drainage (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The original protocol required 50 subjects that completed 5 days of treatment. With protocol amendment 2, the criteria for enrollment/completion was reduced to 1 day of treatment. Subjects were required to have a minimum of 3 IV APAP doses per day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may publish 18 months after Cadence's final evaluation of all study data from all sites, whichever occurs first.Manuscripts/abstracts will be provided to Cadence for review and comment at least 30 days prior to submission.Cadence shall have 30 days to respond with comments.